CLINICAL TRIAL: NCT03151720
Title: A Single-Dose, Randomized, Open-Label, Two-Treatment, Four-Period, Crossover Study to Assess the Relative Bioavailability of Xisimin (Loratadine) Tablets Under Fasting and Fed Conditions in Healthy Subjects Compared to Clarityne Tablets
Brief Title: A Study to Assess the Relative Bioavailability of Xisimin (Loratadine) Tablets Under Fasting and Fed Conditions in Healthy Participants Compared to Clarityne Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108321; 1754415ALY1001 (Other: Xian-Janssen Pharmaceutical Ltd., China)
Record Dates: First submitted 2017-04-28; First posted 2017-05-12 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Healthy
MeSH Terms: interventions — Loratadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Sequence 1 (ABAB) (Experimental): Participants will receive 10 milligram (mg) loratadine (1*10 mg oral tablet) as Xisimin (Treatment A) on Day 1 of Period 1 and Period 3 and 10 mg loratadine (1*10 mg oral tablet) administered as Clarityne (Treatment B) on Day 1 of Period 2 and Period 4 under fasted condition. A washout period of at least 7 days will be maintained between each treatment administration.
  Interventions: Drug: loratadine (Xisimin [Test Treatment]); Drug: loratadine (Clarityne [Reference Treatment])
- Cohort 1: Sequence 2 (BABA) (Experimental): Participants will receive Treatment B on Day 1 of Period 1 and Period 3 and Treatment A on Day 1 of Period 2 and Period 4 under fasted condition. A washout period of at least 7 days will be maintained between each treatment administration.
  Interventions: Drug: loratadine (Xisimin [Test Treatment]); Drug: loratadine (Clarityne [Reference Treatment])
- Cohort 2: Sequence 1 (ABAB) (Experimental): Participants will receive Treatment A on Day 1 of Period 1 and Period 3 and Treatment B on Day 1 of Period 2 and Period 4 under fed condition. A washout period of at least 7 days will be maintained between each treatment administration.
  Interventions: Drug: loratadine (Xisimin [Test Treatment]); Drug: loratadine (Clarityne [Reference Treatment])
- Cohort 2: Sequence 1 (BABA) (Experimental): Participants will receive Treatment B on Day 1 of Period 1 and Period 3 and Treatment A on Day 1 of Period 2 and Period 4 under fed condition. A washout period of at least 7 days will be maintained between each treatment administration.
  Interventions: Drug: loratadine (Xisimin [Test Treatment]); Drug: loratadine (Clarityne [Reference Treatment])

INTERVENTIONS:
Drug: loratadine (Xisimin [Test Treatment]) — Participants will receive 10 mg loratadine as Xisimin (test treatment) as per the treatment sequence.
  Other Names: JNJ-1754415-AAA
Drug: loratadine (Clarityne [Reference Treatment]) — Participants will receive 10 mg loratadine as Clarityne (reference treatment) as per the treatment sequence.

SUMMARY:
The purpose of this study is to establish the relative bioavailability of Xisimin (loratadine) compared to Clarityne in healthy participants receiving a single dose of 10 milligram (mg) under fasting condition as part of Cohort 1 and under fed condition as part of Cohort 2.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI, weight [kilogram]/height^2 [meter^2]) between 19.0 and 26.0 kg/m2 (kilogram per meter square) (inclusive); body weight of male participants not less than 50 kilogram (kg) and body weight of female participants not less than 45 kg
* If a woman, must be surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control (example, prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before entry, throughout the study, and for 1 month after the last dose of study drug
* If a woman, must have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day -1 of each treatment period
* If a woman, must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 2 months after receiving the last dose of study drug
* If a man who is sexually active with a woman of childbearing potential and has not had a vasectomy, must agree to use an adequate contraception method as deemed appropriate by the investigator (example, vasectomy, double-barrier, partner using effective contraception) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug. Must agree to continue using an appropriate method of birth control during the study and for 3 month after the last dose of study drug

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), gastrointestinal disease, lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or on Day -1 of each treatment period as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs or 12 lead electrocardiogram (ECG) at screening or on Day -1 of each treatment period as deemed appropriate by the investigator
* Clinically significant abnormal chest radiography at screening as deemed appropriate by the investigator
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for oral contraceptives and paracetamol within 14 days before the first dose of the study drug is scheduled

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-07-08 (Actual); Study Completion 2017-07-08 (Actual)

PRIMARY OUTCOMES:
Relative Bioavailability of Xisimin Compared With Clarityne | Cohort 1 and Cohort 2: Predose, 0.25 hour (h), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, 24h, 48h, 72h, 96h postdose
  Bioavailability means the extent to which the active ingredient of a drug dosage form becomes available at the site of drug action or in a biological medium believed to reflect accessibility to a site of action. Relative bioavailability is the percentage of the administered dose that is systemically available, calculated as: (AUC [0-infinity] of test divided by AUC [0-infinity] of reference) multiplied by 100, where the reference treatment is a non-intravenous administration.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Loratadine | Cohort 1 and Cohort 2: Predose, 0.25h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, 24h, 48h, 72h, 96h postdose
  The Cmax is the maximum observed plasma concentration.
Area Under the Plasma Concentration-time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) for Loratadine | Cohort 1 and Cohort 2: Predose, 0.25h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, 24h, 48h, 72h, 96h postdose
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-time Curve From Time Zero to Infinite Time (AUC[0-infinity]) for Loratadine | Cohort 1 and Cohort 2: Predose, 0.25h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, 24h, 48h, 72h, 96h postdose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Number of Participants With Adverse Events (AE) as a Measure of Safety and Tolerability | From Screening to Day 5 of Period 4 (Approximately 54 days)
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (1):
- Tri-Service Genaral Hospital, Taipei, Taiwan